CLINICAL TRIAL: NCT00564655
Title: Regional Anesthesia Block of the Transversus Abdominis Plane in Children Undergoing Gastric Tube Insertion
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000011192
Record Dates: First submitted 2007-11-27; First posted 2007-11-28 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Anesthesia; Enteral Nutrition
Keywords: pediatrics; Gastric Tube Insertion; Anesthesia; Regional Anesthetic; Transversus Abdominal Plane
MeSH Terms: interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients in the control group will receive localized infiltration of local anesthesia at the beginning of the procedure as is current standard practice.
  Interventions: Procedure: bupivacaine with epinephrine (mid and upper abdomen)
- 2 (Experimental): Patients in the experimental group will receive a regional anesthetic blockade of the anterior abdominal wall via the transversus abdominis plane.
  Interventions: Procedure: bupivacaine with epinephrine (transversus abdominis plane)

INTERVENTIONS:
Procedure: bupivacaine with epinephrine (mid and upper abdomen) — Patients will receive localized infiltration of local anesthesia (0.25% bupivacaine with epinephrine 1:200,000) at the beginning of the procedure as is current standard practice. Localized anaesthetic of the mid and upper abdomen.
  Arms: 1
Procedure: bupivacaine with epinephrine (transversus abdominis plane) — 0.6 cc/kg (to a maximum of 20 ccs) of 0.25% bupivacaine with epinephrine 1:200,000 will be injected into the neuro-vascular plane between the internal oblique and transversus abdominis muscles. Regional anaesthetic block of the transversus abdominis plane.
  Arms: 2

SUMMARY:
The objective of this trial is to examine if regional anesthetic blockade of the anterior abdominal wall via the transversus abdominis plane is a safe and feasible method of providing analgesia for children undergoing gastric tube insertion.

DETAILED DESCRIPTION:
Regional abdominal field blockade has been demonstrated to deliver effective analgesia for procedures involving the anterior abdominal wall and may represent a feasible, minimally invasive alternative to central neuraxial blockade for some procedures and surgery of the abdomen.

Regional anesthesia and analgesia techniques are commonly advocated for post-operative pain control in pediatric surgical practice. Regional techniques decrease morphine requirements and improve the quality of post-operative pain control and patient-parent satisfaction. The most commonly used technique is caudal anesthesia, which is generally indicated for urologic surgery, inguinal hernia repair and lower extremity surgery. Complications are rare and usually minor, however, the caudal technique is limited in its ability to provide reliable analgesia to the abdominal wall and for surgical procedures involving the mid and upper abdomen. A reasonable alternative for these surgical procedures is to perform a formal lumbar epidural. This provides excellent post-operative analgesia and complications are rare. However, when complications do occur they are not minor. Because of the risks and potential complications of epidural catheter insertion, current clinical experience reveals an unwillingness for parents to consent to this technique.

On average, two hundred gastric tube insertions are performed in Image Guided Therapy (IGT) per annum (year) in this institution. Current standard practice for post-procedure pain control is local infiltration of the insertion site with local anesthetic during the procedure and intravenous morphine supplemented by rectal acetaminophen post-operatively. A retrospective review of this patient group demonstrates that approximately 80% of patients require one to three doses of morphine in the first 12 - 16 hours after the procedure. Even a single dose of intravenous morphine can increase the incidence of vomiting in children undergoing day surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - III
* One to ten years of age
* Scheduled to undergo gastric tube insertion in IGT
* Signed informed consent

Exclusion Criteria:

* Patients requiring emergency procedures
* Refusal of regional block
* History of seizure disorder
* Allergy or sensitivity to bupivacaine, morphine, or radiological contrast
* Hepatic disease
* Bleeding disorder
* Use of pre-operative sedation
* Skin lesions or wounds at site of proposed needle insertion
* Evidence of peritonitis or septicemia
* Patients with ventriculo-peritoneal shunts in situ
* Patients taking any of the following drugs: procainamide, disopyramide, flecainide, mexiletine, cimetidine and ranitidine

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2007-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | For 24 hours after the time of first eye-opening post-procedure
Pain, sedation, nausea & vomiting scores | Pre-procedure; every 15 minutes from time of first eye-opening post-procedure until discharge from post-anesthesia care unit (PACU); on the ward at 2, 4, 8, 12, 16, and 24 hours

SECONDARY OUTCOMES:
Time until the patient is discharged from PACU to the ward | At time of PACU discharge
Parent satisfaction with analgesia and the procedure | On the day following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Conor Mc Donnell, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada